CLINICAL TRIAL: NCT01441245
Title: Continuous Versus Intermittent Loop Diuretics Infusion Dosing in Acute Heart Failure: Effects on Renal Function, Outcome and BNP Levels
Brief Title: Loop Diuretics Administration and Acute Heart Failure
Acronym: diurHF
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Siena (Other)
Responsible Party: Principal Investigator, Alberto Palazzuoli MD PhD, Consultant cardiologist, University of Siena
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: diuretic1
Record Dates: First submitted 2011-09-22; First posted 2011-09-27 (Estimated); Results first posted 2016-02-02 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2017-12

CONDITIONS: Acute Heart Failure
Keywords: acute heart failure; diuretics; BNP; Renal function; acute decompensated Heart Failure,; volume overload
MeSH Terms: conditions — Edema

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Continuous furosemide infusion (Experimental): The group that received the continuous infusion of furosemide (cIV), consisted of 30 patients;
  Interventions: Drug: furosemide infusion
- Intermittent furosemide infusion (Experimental): The group that received the bolus infusion of furosemide (iIV), consisted of 27 patients
  Interventions: Drug: furosemide infusion

INTERVENTIONS:
Drug: furosemide infusion — Patients were randomized in a 1:1 ratio to receive furosemide dose divided into twice-daily bolus injection (group 0) or continuous infusion (group 1)(mixed as a 1:1 ratio in 5% dextrose in water) for a time period ranging from 72 to 120 hours. The mean daily diuretic dosage was similar in the two groups. The median time from presentation to randomization was 16 hours, and the median duration of study-drug administration was 112± 24 hours
  Other Names: Continuous vs intermittent intravenous furosemide infusion

SUMMARY:
Intravenous loop diuretics is the therapy most commonly used to treat pulmonary congestion and systemic fluid overload. In theory, continuous infusion should allow for a more consistent diuresis, avoiding the sodium reabsorption in the distal tubule as well as the neurohormonal activation. This should lead to renal function improvement and BNP decrease.

DETAILED DESCRIPTION:
Patients were eligible if they were admitted with a primary diagnosis of ADHF, randomized within 12 h after hospital presentation, and with evidence of volume overload (pulmonary congestion) on a chest X-ray study and had BNP levels >100 pg/ml. Patients also displayed mild to moderate renal dysfunction with creatinine values up to 1.4 mg/dl. Some patients were supported with non invasive ventilation before randomization. Once the initial 12 h dose was determined, patients were randomized using a 1:1 ratio using a computer-generated scheme to receive the furosemide dose either divided into a twice-daily bolus injection or in a continuous infusion (mixed as a 1:1 ratio in 5 % dextrose in water) for a time period ranging from 72 to 120 h. The randomization was casual, and the physicians did not previously know the assigned arm. The dose escalation and subsequent titration of furosemide was guided by clinical response in terms of urine output volume and body weight reduction .Before randomization, renal function parameters and BNP levels were measured in all patients. Subsequent titration of the furosemide dosage was at the discretion of the attending physician, but was guided by a dose-escalation algorithm based on the treatment response (weight loss and urine output volume), symptom improvement, changes in renal function, electrolyte balance, and chest radiography. The specific doses of furosemide and the use of additional agents to manage ADHF (dopamine, IV vasodilators, hypertonic saline infusion) were decided based upon blood pressure measurements, renal function evaluation and diuresis response. Supplementary treatment was left to the discretion of the treating physician. The duration of infusion was continued for up to 72 h, at 48 h the physicians had the possibility to adjust diuretic dose administration on the basis of the clinical response. After 72 h the treatment could be stopped or continued for an additional 36-48 h depending on the patient's condition and diuresis response. Acute kidney injury (AKI) was defined following the RIFLE criteria.

Abbreviations:

(AKI) Acute kidney injury (ADHF) Acute decompensated heart failure (BNP) B-type natriuretic peptide (CHD) Coronary heart disease (cIV) Continuous infusion (iIV) Intermittent infusione (eGFR)Estimated glomerular filtration rate (Hb) Hemoglobin (HF) Heart failure (Hct) Hematocrit (LVEF) Left ventricular ejection fraction (RBC) Red blood cells

ELIGIBILITY:
Inclusion Criteria:

* Patients took part in the random sample selection if they met the diagnostic criteria for acute decompensated HF.
* Patients with primary diagnosis of ADHF, volume overload with cardia dilation and LVEF <50%, and had BNP levels >100 pg/ml.

Exclusion Criteria:

* Patients were excluded if they had received more than 2 IV doses of furosemide or any continuous infusion of furosemide 1 month before randomization
* If they had end-stage renal disease or the need for renal replacement therapy, isolated diastolic dysfunction.
* Recent myocardial infarction

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2010-04 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2017-12-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Palazzuoli, MD, Principal Investigator — Department of Internal Medicine, Cardiology Unit, Le Scotte Hospital, Siena
Locations (1):
- Department of Internal Medicine, Cardiology Section Center, Siena, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Palazzuoli A, Pellegrini M, Franci B, Beltrami M, Ruocco G, Gonnelli S, Angelini GD, Nuti R. Short and long-term effects of continuous versus intermittent loop diuretics treatment in acute heart failure with renal dysfunction. Intern Emerg Med. 2015 Feb;10(1):41-9. doi: 10.1007/s11739-014-1112-5. Epub 2014 Aug 3. PMID 25087085
- [Result] Felker GM, Lee KL, Bull DA, Redfield MM, Stevenson LW, Goldsmith SR, LeWinter MM, Deswal A, Rouleau JL, Ofili EO, Anstrom KJ, Hernandez AF, McNulty SE, Velazquez EJ, Kfoury AG, Chen HH, Givertz MM, Semigran MJ, Bart BA, Mascette AM, Braunwald E, O'Connor CM; NHLBI Heart Failure Clinical Research Network. Diuretic strategies in patients with acute decompensated heart failure. N Engl J Med. 2011 Mar 3;364(9):797-805. doi: 10.1056/NEJMoa1005419. PMID 21366472
- [Derived] Ruocco G, Feola M, Nuti R, Luschi L, Evangelista I, Palazzuoli A. Loop Diuretic Administration in Patients with Acute Heart Failure and Reduced Systolic Function: Effects of Different Intravenous Diuretic Doses and Diuretic Response Measurements. J Clin Med. 2019 Nov 2;8(11):1854. doi: 10.3390/jcm8111854. PMID 31684094
- [Derived] Ruocco G, Evangelista I, Franci B, Lucani B, Martini S, Nuti R, Palazzuoli A. Combination of ST2 and B-type natriuretic peptide in diabetic patients with acute heart failure: relation with ventricular stiffness and outcome. J Cardiovasc Med (Hagerstown). 2019 Feb;20(2):81-90. doi: 10.2459/JCM.0000000000000741. PMID 30540645
- [Derived] Palazzuoli A, Pellegrini M, Ruocco G, Martini G, Franci B, Campagna MS, Gilleman M, Nuti R, McCullough PA, Ronco C. Continuous versus bolus intermittent loop diuretic infusion in acutely decompensated heart failure: a prospective randomized trial. Crit Care. 2014 Jun 28;18(3):R134. doi: 10.1186/cc13952. PMID 24974232

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Department of Internal Medicine, Cardiology Section Centre into a Para-Intensive Unit (Siena, Italy) from April 2011 to December 2012.
Pre-assignment Details: 22 were excluded because of normal renal function at baseline, 11 for receiving different dosages of intravenous furosemide, 4 for isolated diastolic HF
Groups:
- cIV Group: The group that received the continuous infusion of furosemide (cIV), consisted of 30 patients.
- iIV Group: The second group that received the same drug in bolus injections twice a day (iIV), consisted of 27 patients.
Period: Overall Study
Arm/Group | cIV Group | iIV Group
Started | 30 | 27
Completed | 30 | 27
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- iIV Group: The group that received the intermittent infusion of furosemide (iIV), consisted of 27 patients.
- Total: Total of all reporting groups
Arm/Group | cIV Group | iIV Group | Total
Number analyzed (Participants) | 30 | 27 | 57
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 6 | 11
  >=65 years | 25 | 21 | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 71 (7) | 73 (8) | 72 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 13 | 27
  Male | 16 | 14 | 30
Region of Enrollment [Number; unit: participants]
  Italy | 30 | 27 | 57

OUTCOME MEASURES:

1. Primary Outcome: Evaluation of Mean Urine Output Volume During the Infusion Period
Description: this study aimed to evaluate the effects of continuous infusion of furosemide in comparison to twice daily regimens at similar doses with respect to changes in renal function in terms of creatinine levels and GFR, urine output and BNP levels from admission to discharge
Time Frame: time period ranging from 72 h to 120 h.
Measure: Mean (Standard Deviation); unit: mL
Groups:
- Urine Output in cIV; Urine Output in iIV: Evaluation of urine output in Intermittent intravenous furosemide infusion group
Arm/Group | Urine Output in cIV | Urine Output in iIV
Number analyzed (Participants) | 30 | 27
mL | 2505 (796) | 2140 (468)
Statistical Analysis 1: Comparison: Urine Output in cIV vs Urine Output in iIV; Continuous variables are expressed as mean ± standard deviation (SD) and compared with t test for independent groups. p values <0.05 were considered significant; Test type: Non-Inferiority or Equivalence — The sample size used was preliminarily calculated from each co-primary endpoint. We included the following assumptions: (1) a 30 % or more effect size in the difference between mean paired changes in continuous co-primary endpoints (eGFR, creatinine, BNP and diuresis); standard variation of each group data not exceeding 20 %; (2) alpha = 0.05 two-tailed and (3) power (1-beta) = 80 %; p = 0.04, t-test, 2 sided

2. Secondary Outcome: Length of Hospitalization in the Two Groups
Description: percentage of participants with hospital stay > 10 days
Time Frame: in-hospital
Population: Qualitative variables are expressed as percentage and compared with chi-square test . p values <0.05 were considered significant.
Measure: Number; unit: percentage of partecipants
Groups:
- Lenght of Hospitalization in cIV: Prevalence of hospital stay > 10 days in continuous intravenous furosemide infusion.
- Lenght of Hospitalization in iIV: Prevalence of hospital stay > 10 days in intermittent intravenous furosemide infusion.
Arm/Group | Lenght of Hospitalization in cIV | Lenght of Hospitalization in iIV
Number analyzed (Participants) | 30 | 27
percentage of partecipants | 80 | 44
Statistical Analysis 1: Comparison: Lenght of Hospitalization in cIV vs Lenght of Hospitalization in iIV; Qualitative variables are expressed as percentage and compared with chi-square test. p values <0.05 were considered significant; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.01, Chi-squared

3. Primary Outcome: Evaluation of Renal Function in Terms of Creatinine Levels at Discharge
Time Frame: from admission to discharge, an average of 12 days
Population: All data were analyzed with intention-to-treat. Continuous variables are expressed as mean ± standard deviation (SD) and compared with t test for independent groups. p values <0.05 were considered significant.
Measure: Mean (Standard Deviation); unit: mg/dL
Groups:
- Creatinine at Discharge in cIV: Mean creatinine at discharge in continuous intravenous fursoemide infusion.
- Creatinine at Discharge in iIV: Mean creatinine at discharge in intermittent intravenous fursoemide infusion.
Arm/Group | Creatinine at Discharge in cIV | Creatinine at Discharge in iIV
Number analyzed (Participants) | 30 | 27
mg/dL | 1.78 (0.5) | 1.51 (0.3)
Statistical Analysis 1: Comparison: Creatinine at Discharge in cIV vs Creatinine at Discharge in iIV; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.01, t-test, 2 sided

4. Primary Outcome: Evaluation of Renal Function in Terms of Changes in Creatinine Levels
Description: evaluation of renal function in terms of changes in creatinine levels during hospitalization in the two arms.
Time Frame: participants were followed for the duration of hospital stay, an average of 13 days
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mg/dL
Groups:
- Changes in Creatinine in cIV Group: The group that received the continuous infusion of furosemide (cIV), consisted of 30 patients
  furosemide infusion: Patients were randomized in a 1:1 ratio to receive furosemide dose divided into twice-daily bolus injection (group 0) or continuous infusion (group 1)(mixed as a 1:1 ratio in 5% dextrose in water) for a time period ranging from 72 to 120 hours. The mean daily diuretic dosage was similar in the two groups. The median time from presentation to randomization was 16 hours, and the median duration of study-drug administration was 112± 24 hours
- Changes in Creatinine in iIV Group: The group that received the bolus infusion of furosemide (iIV), consisted of 27 patients
  furosemide infusion: Patients were randomized in a 1:1 ratio to receive furosemide dose divided into twice-daily bolus injection (group 0) or continuous infusion (group 1)(mixed as a 1:1 ratio in 5% dextrose in water) for a time period ranging from 72 to 120 hours. The mean daily diuretic dosage was similar in the two groups. The median time from presentation to randomization was 16 hours, and the median duration of study-drug administration was 112± 24 hours
Arm/Group | Changes in Creatinine in cIV Group | Changes in Creatinine in iIV Group
Number analyzed (Participants) | 30 | 27
mg/dL | -0.10 (0.30) | -0.50 (0.34)
Statistical Analysis 1: Comparison: Changes in Creatinine in cIV Group vs Changes in Creatinine in iIV Group; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.02, t-test, 2 sided

5. Primary Outcome: Evaluation of B-type Natriuretic Peptide (BNP) Levels From Admission to the End of Treatment
Time Frame: from admission to discharge, an average of 12 days
Measure: Mean (Standard Deviation); unit: pg/ml
Groups:
- BNP Levels at Discharge in cIV Group: The group that received the continuous infusion of furosemide (cIV), consisted of 30 patients
  furosemide infusion: Patients were randomized in a 1:1 ratio to receive furosemide dose divided into twice-daily bolus injection (group 0) or continuous infusion (group 1)(mixed as a 1:1 ratio in 5% dextrose in water) for a time period ranging from 72 to 120 hours. The mean daily diuretic dosage was similar in the two groups. The median time from presentation to randomization was 16 hours, and the median duration of study-drug administration was 112± 24 hours
- BNP Levels at Discharge in iIV Group: The group that received the bolus infusion of furosemide (iIV), consisted of 27 patients
  furosemide infusion: Patients were randomized in a 1:1 ratio to receive furosemide dose divided into twice-daily bolus injection (group 0) or continuous infusion (group 1)(mixed as a 1:1 ratio in 5% dextrose in water) for a time period ranging from 72 to 120 hours. The mean daily diuretic dosage was similar in the two groups. The median time from presentation to randomization was 16 hours, and the median duration of study-drug administration was 112± 24 hours
Arm/Group | BNP Levels at Discharge in cIV Group | BNP Levels at Discharge in iIV Group
Number analyzed (Participants) | 30 | 27
pg/ml | 679 (397) | 949 (548)
Statistical Analysis 1: Comparison: BNP Levels at Discharge in cIV Group vs BNP Levels at Discharge in iIV Group; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.04, t-test, 2 sided
Statistical Analysis 2: Comparison: BNP Levels at Discharge in cIV Group vs BNP Levels at Discharge in iIV Group; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.01, Regression, Linear; Risk Ratio (RR) = 2.06, 95% CI 2-sided [1.65 to 2.57] — BNP levels at discharge >500 pg/ml (RR: 2.06 [1.65-2.57];)

6. Primary Outcome: Change in Brain Natriuretic Peptide (BNP) Levels From Admission to the Discharge
Time Frame: participants were followed for the duration of hospital stay, an average of 13 days
Population: Continuous variables are expressed as mean ± standard deviation (SD) and compared with t test for independent groups. p values <0.05 were considered significant.
Measure: Mean (Standard Deviation); unit: pg/mL
Groups:
- BNP Change in cIV; BNP Change in iIV: Evaluation of BNP change in Intermittent intravenous furosemide infusion group
Arm/Group | BNP Change in cIV | BNP Change in iIV
Number analyzed (Participants) | 30 | 27
pg/mL | -525 (615) | -148 (463)
Statistical Analysis 1: Comparison: BNP Change in cIV vs BNP Change in iIV; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.03, t-test, 2 sided

7. Primary Outcome: Evaluation of Renal Function in Terms of Changes in GFR
Time Frame: from admission to discharge, an average of 12 days
Measure: Mean (Standard Deviation); unit: (ml/min·1.73 m2)
Groups:
- GFR Change in cIV: Mean GFR change in continuous intravenous fursoemide infusion.
- GFR Change in iIV: Mean GFR change in intermittent intravenous fursoemide infusion.
Arm/Group | GFR Change in cIV | GFR Change in iIV
Number analyzed (Participants) | 30 | 27
(ml/min·1.73 m2) | -3.18 (2.45) | -1.93 (2.90)
Statistical Analysis 1: Comparison: GFR Change in cIV vs GFR Change in iIV; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.01, t-test, 2 sided

8. Primary Outcome: Evaluation of Renal Function in Terms of GFR Values at Discharge
Time Frame: from admission to discharge, an average of 12 days
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: (ml/min·1.73 m2)
Groups:
- GFR at Discharge in cIV: Mean GFR at discharge in continuous intravenous fursoemide infusion.
- GFR at Discharge in iIV: Mean GFR at discharge in intermittent intravenous fursoemide infusion.
Arm/Group | GFR at Discharge in cIV | GFR at Discharge in iIV
Number analyzed (Participants) | 30 | 27
(ml/min·1.73 m2) | 44.8 (6.1) | 46.7 (6.1)
Statistical Analysis 1: Comparison: GFR at Discharge in cIV vs GFR at Discharge in iIV; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.05, t-test, 2 sided

9. Secondary Outcome: Dopamine Infusion During Hospitalization
Time Frame: in-hospital
Measure: Number; unit: percentage of partecipants
Groups:
- Dopamine Infusion in cIV: Prevalence of dopamine infusion in continuous intravenous furosemide infusion.
- Dopamine Infusion in iIV: Prevalence of dopamine infusion in intermittent intravenous furosemide infusion.
Arm/Group | Dopamine Infusion in cIV | Dopamine Infusion in iIV
Number analyzed (Participants) | 30 | 27
percentage of partecipants | 50 | 26
Statistical Analysis 1: Comparison: Dopamine Infusion in cIV vs Dopamine Infusion in iIV; Qualitative variables are expressed as percentage of partecipants and compared with chi-square test. p-value equal or lower than 0.05 are considered statistically significant; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.01, Chi-squared

ADVERSE EVENTS:
Time Frame: The 6-months follow-up events encompassed: cardiac death, rehospitalization for all cardiovascular causes, and severe renal insufficiency needing hemodialysis.
Arm/Group | cIV Group | iIV Group
Serious Adverse Events (participants affected / at risk) | 14/30 | 9/27
Other Adverse Events (participants affected / at risk) | 0/30 | 0/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | cIV Group (N=30) | iIV Group (N=27)
death (Cardiac disorders) | 6 (6) | 3 (3) — Cardiac death
rehospitalization for all cardiovascular causes (Cardiac disorders) | 8 (8) | 6 (6)
needing renal replacement therapy (Renal and urinary disorders) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Our study didn't explain the reasons of renal dysfunction during treatment. Concurrent evaluation of BUN could further clarify the primary defect.The multivariate analysis could be inadequate for small sample; we intend to continue enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No